CLINICAL TRIAL: NCT02256423
Title: A Single-dose, Randomised, Crossover Study to Compare the Pharmacokinetics of Three Formulations of Ibuprofen in Healthy Fasting Male and Female Subjects
Brief Title: A Study Comparing Three Formulations of Ibuprofen in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Simbec Research (Industry)
Responsible Party: Principal Investigator, Girish Sharma, Associate Medical Director, Simbec Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RD 680/25772
Record Dates: First submitted 2014-09-16; First posted 2014-10-03 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-09

CONDITIONS: Healthy Volunteer Study
Keywords: Ibuprofen; healthy volunteer study; pharmacokinetics
MeSH Terms: interventions — Tablets; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- REFERENCE 1: Nurofen® 200 mg tablet (Active Comparator): Single group 3-way crossover study
  Interventions: Drug: REFERENCE 1: Nurofen® 200 mg tablet
- REFERENCE 2: Ibuprofen 200 mg soft gel capsule (Active Comparator): Single group 3-way crossover study
  Interventions: Drug: REFERENCE 2: Ibuprofen 200 mg soft gel capsule
- ibuprofen 200 mg soft gel capsule (Experimental): single group, 3-way cross
  Interventions: Drug: ibuprofen 200 mg soft gel capsule

INTERVENTIONS:
Drug: REFERENCE 1: Nurofen® 200 mg tablet
  Arms: REFERENCE 1: Nurofen® 200 mg tablet
Drug: REFERENCE 2: Ibuprofen 200 mg soft gel capsule
  Arms: REFERENCE 2: Ibuprofen 200 mg soft gel capsule
Drug: ibuprofen 200 mg soft gel capsule
  Arms: ibuprofen 200 mg soft gel capsule

SUMMARY:
This is an open-label, randomised, 3-period, 3-sequence single-dose crossover study to determine the comparative pharmacokinetic profile of the Test Investigational Medicinal Product (IMP) Ibuprofen 200 mg soft gel capsule (lipid formulation) with that from the reference products Nurofen® 200 mg tablet and ibuprofen 200 mg soft gel capsule following single dose administration in healthy male and female subjects.

The study comprises of a pre-study screen (within 14 days of the first dose), followed by 3 Treatment Periods (1, 2 and 3) and a post study follow up (3 - 7 days after the last dose). Each Treatment Period is of 1 day in duration, from the afternoon before dosing (Day -1) until 12 hours (h) post-dose (Evening of Day 1). Study drug is administered on the morning of Day 1 following an overnight fast. PK samples will be collected pre-dose and up to 12 h post-dose (x15 samples) for the measurement of ibuprofen. Safety is evaluated at specified times throughout the study. There is at least 48 h between dose administrations.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females between 18 and 50 years of age.
2. Female subject of child bearing potential with a negative pregnancy test at the Screening Visit and willing to use an effective method of contraception if applicable (unless of non-childbearing potential or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from Day 1 until 3 months afterwards.
3. Female subject of non-child bearing potential with negative pregnancy test at the Screening Visit. For the purposes of this study, this is defined as the subject being amenorrheic for at least 12 consecutive months or at least 4 months post-surgical sterilisation (including bilateral fallopian tube ligation or bilateral oophorectomy with or without hysterectomy). Menopausal status will be confirmed by demonstrating at screening that levels of follicle stimulating hormone (FSH) fall within the respective pathology reference range. In the event a subject's menopause status has been clearly established (for example, the subject indicates she has been amenorrheic for 10 years), but FSH levels are not consistent with a post-menopausal condition, determination of subject eligibility will be at the discretion of the Chief Investigator following consultation with the Sponsor's Responsible Physician.
4. Subject with a Body Mass Index (BMI) of 18-30 kilogram (kg)/metre square (m2). Body Mass Index = Body weight in kg / [Height in m]2.
5. Subject with no clinically significant abnormal serum biochemistry, haematology and urine examination values within 14 days of the first dose.
6. Subject with a negative urinary drugs of abuse screen, determined within 14 days of the first dose (a positive alcohol result may be repeated at the discretion of the Investigator).
7. Subject with negative human immunodeficiency virus (HIV), hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
8. Subject with no clinically significant abnormalities in 12-lead ECG determined within 14 days of the first dose.
9. Subject must be available to complete the study (including all follow up visits) and comply with study restrictions.
10. Subject must satisfy a medical examiner about their fitness to participate in the study.
11. Subject must provide written informed consent to participate in the study.

Exclusion Criteria:

1. History of allergy to NSAIDs or aspirin and history of peptic ulcer or gastrointestinal bleeding.
2. A clinically significant history of gastrointestinal disorder likely to influence drug absorption, such as Gastroesophageal reflux disease
3. Receipt of regular medication within 14 days of the first dose that may have an impact on the safety and objectives of the study (at the Investigator's discretion).
4. Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
5. A clinically significant history of previous allergy / sensitivity to ibuprofen.
6. A clinically significant history of drug or alcohol abuse.
7. Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
8. Participation in a New Chemical Entity clinical study within the previous 4 months or a marketed drug clinical study within the previous 3 months. (N.B. washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
9. Donation of 450 mL or more blood within the previous 3 months.
10. Subjects who are current smokers, or those who have used nicotine products within the previous 3 months.
11. Subject with positive human immunodeficiency virus (HIV), hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
12. Any subject who, in the judgment of the Investigator, is likely to be non-compliant with study procedures and/or restrictions during the study, or unable to cooperate because of a language problem or poor mental development.
13. Subjects must not have taken over the counter drugs and herbal remedies and supplements should not be taken from 7 days prior to the first dose and throughout the duration of the study dosing periods.
14. Prescribed drugs should not be taken for 7 days before the first dose and throughout the duration of the study dosing periods. This does not include the oral contraceptive pill.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | PK samples are taken up to 12 hours of each study period.
  Maximum plasma concentration (Cmax), time to Cmax (tmax), elimination rate constant (λz), terminal half-life (t1/2), area under the concentration-time curve (AUC) from time of dosing to last measurable concentration (AUC0-t), partial area under plasma concentration time curve at the following nominal blood sampling time points 15min, 30min, 45min, 1h, 1.20h, 1.40h and 2h (AU0-n), AUC extrapolated to infinity (AUC0-∞), plasma clearance (CL/F), MRT (mean residence time) and AUC% extrapolated (residual area).

SECONDARY OUTCOMES:
Safety | participants will be followed for the duration of stay, an expected average of 3 weeks
  AEs, vital signs (sitting blood pressure and pulse), ECG (heart rate, PR interval, QRS width, QT interval and QTcB interval) and laboratory (haematology, biochemistry and urinalysis) data.

CONTACTS AND LOCATIONS:
Overall Officials: Girish Sharma, MBBS, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Limited, Merthyr Tydfil, United Kingdom